CLINICAL TRIAL: NCT00744107
Title: The Cobra II Study: Use of the Cobra™ Cobalt Super Alloy Coronary Stent System in the Treatment of Coronary Artery Disease
Brief Title: Cobra II Study: Use of the Cobra™ Cobalt Super Alloy Coronary Stent System in the Treatment of Coronary Artery Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medlogics Device Corporation (Industry)
Collaborators: Baim Institute for Clinical Research (Other); Stanford University (Other)
Responsible Party: Medlogics Device Corporation, Medlogics Device Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59-2004
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Artery Disease
Keywords: Ischemic coronary artery disease in native coronary arteries; Single stent; RVD 2.5- 4.0mm; Lesion length up to 26mm; de novo or previously unstented lesions
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: PCI with the Cobra™ Cobalt Super Alloy Coronary Stent System — stent placement, single-arm study

SUMMARY:
To demonstrate the safety and efficacy of the Cobra Cobalt Super Alloy Balloon-Expandable Coronary Stent System for the treatment of de novo and restenotic (previously unstented) lesions in native coronary arteries in subjects with coronary artery disease (CAD) having a reference vessel diameter (RVD) between 2.5 - 4.0 mm and a lesion length ≤ 26 mm amenable to percutaneous coronary intervention (PCI) with a single stent in subjects with symptomatic ischemic heart disease.

DETAILED DESCRIPTION:
Safety and Efficacy will be demonstrated by the rate of Target vessel failure (TVF), defined as cardiac death, target vessel myocardial infarction (MI) [Q wave or non-Q wave], or clinically driven target vessel revascularization (TVR) by percutaneous or surgical methods within 270 days of the post-stent placement procedure.

Additionally, Major Adverse Cardiac Events (MACE)at 30, 180 and 270 days defined as a composite of all-cause death, myocardial infarction (MI) (Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion revascularization (TLR) [percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)]will be documented.

ELIGIBILITY:
Inclusion Criteria:

* The subject is ≥ 18 years old;
* Subject is eligible for percutaneous coronary intervention (PCI), stent placement, and emergent coronary artery bypass graft (CABG) surgery;
* Subject has clinical evidence of ischemic heart disease, stable or unstable angina or silent ischemia;
* The subject has a documented left ventricular ejection fraction (LVEF) ≥ 30%;
* The subject or legal representative has been informed of the clinical study and the required follow-up procedures and must provide written informed consent using a form that is reviewed and approved by the Institutional Review Board/Ethics Committee (IRB/EC) for the clinical site;
* Female subjects of childbearing potential must have a negative pregnancy test within 7 days before treatment;
* Subject must agree to comply with the required follow-up procedures (including antiplatelet regimen) to the best of their ability, be geographically available for all study follow-up procedures and visits and not have a known medical condition that precludes completion of the required follow-up visits;
* The lesion is either de novo or restenotic (previously unstented) in nature, located in a native coronary artery AND is ≥ 50% and < 100% stenosed by visual estimate or on-line QCA;
* The target vessel reference diameter ≥ 2.5mm and ≤ 4mm by visual estimate and is appropriate for treatment with available stent diameters of 2.5 mm, to 4.0 mm;
* The lesion length is ≤ 26 mm and able to accommodate placement of a single stent;
* The target lesion is a minimum of 15 mm from any previously placed stent; AND
* The target vessel must have a Thrombolysis In Myocardial Infarction (TIMI) flow ≥ 2

Exclusion Criteria:

* The subject has a known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, ticlopidine and clopidogrel, cobalt, nickel, chromium, molybdenum, or a sensitivity to contrast media, which cannot be adequately pre-medicated;
* A platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a WBC < 3,000 cells/mm³;
* A creatinine level > 2.5 mg/dL within 7 days prior to the index procedure;
* Evidence of an acute myocardial infarction (MI) within 72 hours of the intended treatment (defined as: Q wave (QWMI) or any elevation of creatine kinase myocardial-band (CK-MB) isoenzyme elevated above the Institution's upper limit of normal;
* Any previous PCI (with or without stent) of the target vessel within 30 days prior to the index procedure;
* Previous stent placement anywhere in the target lesion;
* Previous drug eluting stent (DES) deployment anywhere in the target vessel;
* The subject requires staged procedure of any non-target vessel within 30 days post-procedure;
* The subject requires staged procedure of the target vessel within 9 months post-procedure;
* The target lesion requires treatment with a device other than PTCA prior to stent placement (including, but not limited to, cutting balloon, directional coronary atherectomy, excimer laser, rotational atherectomy, thrombectomy, etc.;
* History of a stroke or transient ischemic attack (TIA) within the previous 6 months;
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within the previous 6 months;
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions;
* A known concurrent medical condition resulting in a life expectancy of less than 12 months;
* Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to brachytherapy;
* The subject is currently participating in another investigational device or drug study and has not completed the primary endpoint(s) follow-up phase of that study at least 30 days prior to enrollment in this trial; or interferes with the current trial endpoints; or the subject has previously been enrolled in the study;
* The subject has a known medical condition that will cause them to be non-compliant with the study protocol or confound the data interpretation;
* The target vessel has evidence of thrombus or other lesions having a > 60% stenosis by visual estimate or on-line QCA;
* Target vessel exhibiting multiple lesions with greater than 60% diameter stenosis outside of a range of 5 mm proximal and distal to the target lesion based on visual estimate or on-line QCA;
* The target vessel has evidence (visual or QCA) of excessive tortuosity (two or more 90° bends prior to the target lesion) or is severely calcified; OR
* The target lesion is in an unprotected left main, involves a side branch vessel having a diameter of > 2.0 mm or is at the aorto-ostial location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-07 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF), defined as cardiac death, target vessel myocardial infarction (MI) [Q wave or non-Q wave], or clinically driven target vessel revascularization (TVR) by percutaneous or surgical methods. | 270 days

SECONDARY OUTCOMES:
MACE defined as all-cause death, MI, emergent CABG, or clinically driven TLR; TVF; 6 month In-segment %DS, late lumen loss, binary restenosis and In-stent %DS,late lumen loss, binary restenosis, MLD | 30-, 180- and 270-days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nicolaus J Reifart, PhD, MD, Principal Investigator — Main Taunus Kliniken, Kardiologisches
Locations (7):
- Germany (3):
  - Main Taunus Kliniken, Kardiologisches, Bad Soden
  - St. Vincenz Krankenhaus, Essen
  - Krankenhaus der Barmherzigen Brüder, Trier
- Hadassah Hebrew University Medical Center, Jerusalem, Israel
- Catharina-Ziekenhuis, Eindhoven, Netherlands
- United Kingdom (2):
  - Royal Infirmary, Edinburgh
  - Golden Jubilee Hospital, Glasgow